CLINICAL TRIAL: NCT05256719
Title: a Single-Center, Randomized, Double-Blind, Does-Escalation Phase I Clinical Study to Evaluate the Tolerability, Safety, PK Characteristics of Recombinant Humanized CTLA-4-FC Fusion Protein Injection in Healthy Subjects.
Brief Title: Clinical Study of Recombinant Humanized CTLA-4-FC Fusion Protein Injection in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing VDJBio Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VDJ-002-I
Record Dates: First submitted 2021-12-21; First posted 2022-02-25 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Health Volunteer
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg (Experimental): Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg single dose usage
  Interventions: Biological: Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg
- Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg (Experimental): Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg single dose usage
  Interventions: Biological: Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg
- Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg (Experimental): Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg single dose usage
  Interventions: Biological: Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg
- Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg (Experimental): Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg single dose usage
  Interventions: Biological: Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg
- Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg (Experimental): Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg single dose usage
  Interventions: Biological: Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg
- Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg (Placebo Comparator): Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg , i.v. single dose usage.
  Interventions: Biological: Placebo-1mg/kg
- Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg (Placebo Comparator): Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg, i.v. single dose usage.
  Interventions: Biological: Placebo-2.5mg/kg
- Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg (Placebo Comparator): Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg , i.v. single dose usage.
  Interventions: Biological: Placebo-5mg/kg
- Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg (Placebo Comparator): Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg , i.v. single dose usage.
  Interventions: Biological: Placebo-7.5mg/kg
- Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg (Placebo Comparator): Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg , i.v. single dose usage.
  Interventions: Biological: Placebo-10mg/kg

INTERVENTIONS:
Biological: Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg , i.v. single dose usage.
  Arms: Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg
Biological: Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg , i.v. single dose usage.
  Arms: Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg
Biological: Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg , i.v. single dose usage.
  Arms: Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg
Biological: Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg , i.v. single dose usage.
  Arms: Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg
Biological: Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg , i.v. single dose usage.
  Arms: Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg
Biological: Placebo-1mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg
  Arms: Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 1mg/kg
Biological: Placebo-2.5mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg
  Arms: Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 2.5mg/kg
Biological: Placebo-5mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg
  Arms: Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 5mg/kg
Biological: Placebo-7.5mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg
  Arms: Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 7.5mg/kg
Biological: Placebo-10mg/kg — Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg
  Arms: Placebo Group:Recombinant human CTLA-4-FC fusion protein for injection 10mg/kg

SUMMARY:
This is a single-center, randomized, double-blind, does-escalation Phase I Clinical Study that aim to evaluate the tolerability, safety and PK Characteristics of recombinant humanized CTLA-4-FC fusion protein injection in Healthy Subjects.

DETAILED DESCRIPTION:
This study adopts a single-center,randomized, double-blind, does-escalation, placebo-controlled design.

There are five dose levels of 1mg/kg, 2.5mg/kg, 5mg/kg, 7.5mg/kg and10mg/kg. 2 of 4 subjects in the 1mg/kg dose group receive the test drug and two receive a placebo. 4 of 6 subjects in the 2.5mg/kg dose group receive the test drug and two receive a placebo. 10 of 12 subjects in the 5mg/kg dose group receive the test drug and two receive a placebo. 10 of 12 subjects in the 7.5mg/kg dose group receive the test drug and two receive a placebo. 10 of 12 subjects in the 10mg/kg dose group receive the test drug and two receive a placebo. Subjects are randomly assigned to receive intravenous administration of the test drug or placebo.

The next higher dose group could be initiated only if the stopping rules is not met which are determined by investigator.

ELIGIBILITY:
Inclusion Criteria:

1. For healthy subjects, health was defined as no abnormality or no abnormality of clinical significance during the screening period, such as medical history, physical examination, electrocardiogram, imaging, and laboratory results;
2. Male or female subjects, between 18 and 45 years old (including boundary values);
3. Male subjects should weigh no less than 50.0 kg and female subjects should weigh no less than 45.0 kg. Body mass index (BMI) between 19.0 and 25.0 kg/m2 (including critical value),BMI= weight (kg)/ height 2(m2);
4. Women of reproductive age must use a reliable method of contraception to avoid pregnancy throughout the study period, 4 weeks prior to administration and 3 months after the end of the study, and fertile men must use a reliable method of contraception to avoid pregnancy during the study period and 3 months after the end of the study;
5. Subjects voluntarily participated in the study and signed informed consent.

Exclusion Criteria:

1. Allergic disposition, known or suspected allergy to the test drug or any excipients (disodium hydrogen phosphate and mannitol) or allergy to alcohol/iodine (or iodophor)/ heparin or a history of allergy to any drug, food or pollen, or abnormal serum immunoglobulin E(IgE) tests, conforming to any of these conditions;
2. Have a fertility plan or sperm/egg donation plan during the study period and within 3 months after the study; Female subjects have positive urine/blood pregnancy test at baseline, or are lactating;
3. Female subjects who took oral contraceptives 30 days before and during the trial, or who used long-acting estrogen or progesterone injections or implants 6 months before and during the trial;
4. Patients with central nervous system, cardiovascular system, liver and kidney dysfunction, digestive system, respiratory system and skeletal system diseases (including but not limited to arrhythmia, bradycardia, hypotension, coronary heart disease, bronchial asthma, diabetes, hyperthyroidism, Parkinson's disease, epilepsy, paralysis tremor) Or a history of mental illness and any other diseases or physical conditions that may affect the results of the study;
5. Acute chronic bacterial infection within 3 months before enrollment; At the time of enrollment, any symptoms, signs or abnormal laboratory examination suggested the possibility of acute or subacute infection (such as fever, cough, urination, pain, abdominal pain, diarrhea, skin infection, wound, etc.);
6. Those who had undergone major surgical operations (craniotomy or thoracotomy) within 4 weeks prior to enrollment, or planned to undergo surgery during the study period, and had unhealed wounds, ulcers or fractures;
7. Patients with herpes zoster remission less than 2 months before enrollment;
8. Physical examination or ecg reveals abnormal vital signs: heart rate < 50 beats/min or > 100 times/min (at least 5 minutes after resting), systolic pressure > 140 mmHg or diastolic blood pressure > 90 mmHg, or postural hypotension, body temperature (axillary temperature) 37.3;
9. Blood routine examination: White blood cell (WBC)& LT; 3.0 109 / L or & gt; 9.5 109/L, neutrophils < 1.5 109/L, platelet < 100 109/L; Hemoglobin & Lt; 130g/L(male) or < 110 g/L (women); Bilirubin & gt; 1.2 times normal upper limit, serum creatinine & GT; Upper normal value; AST> Upper limit of normal,ALT> Upper limit of normal;
10. Subjects at risk for tuberculosis (TB) :1) have a history of active TB infection; 2) Tuberculin test positive; 3) Radiological examination indicated past tuberculosis infection;
11. Hiv-ab HCV-AB HBsAg syphilis test results of either positive;
12. Persons with a history of drug or alcohol abuse or positive urine drug screening within 6 months prior to screening;
13. Those who donated blood within 3 months before enrollment or planned to donate blood during the study period and 1 month after the study ended;
14. Patients who had received blood transfusion within 4 weeks prior to enrollment;
15. Subjects who were smokers (who had smoked for more than 6 months prior to screening and smoked more than 5 cigarettes per day), consumed 3 cups of coffee or other caffeine-containing beverages, or 5 cups of tea per day;
16. Prior to screening, use of any prescription over-the-counter drug or herbal medicine with an estimated time of less than 5 half-life of the drug or less than 14 days prior to initial administration, whichever is the longest;
17. Those who received vaccination or immunotherapy within 3 months prior to screening; Those who plan to receive the vaccine during the study period or within 3 months of discontinuing the drug;
18. Patients who cannot tolerate venipunctures and have a history of needle sickness and blood sickness;
19. Participants who participated in any drug clinical trials within 3 months prior to enrollment, or who plan to participate in other drug clinical trials during the study period;
20. The investigator considered that participants were not eligible to participate in the clinical trial for other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by subjects with adverse events | First dose up to last follow-up visit （85 days after administration）
  The number of occurrences and incidence are calculated with vital signs, Electrocardiograms, physical examinations, laboratory tests

SECONDARY OUTCOMES:
Peak concentration (Cmax) | First dose up to last follow-up visit(Day1-Day85）
  Maximum plasma concentration (Cmax) of CTLA-4-FC fusion protein
Peak time (Tmax) | First dose up to last follow-up visit(Day1-Day85）
  Time required to reach peak concentration after administration of CTLA-4-FC fusion protein
Area under the Curve (AUC) | First dose up to last follow-up visit(Day1-Day85）
  Time required to reach peak concentration after administration of CTLA-4-FC fusion protein
Analysis of immunogenicity | First dose up to last follow-up visit（Day1-Day85）
  The number and positive percentage of anti-drug antibody(ADA) and Neutralizing Antibody(NAb) in different dose groups (experimental drug group and placebo group) were calculated

CONTACTS AND LOCATIONS:
Overall Officials: Huiying Rao, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No